CLINICAL TRIAL: NCT06076616
Title: Prehabilitation and Rehabilitation in Breast Cancer Surgery Patients - a Pilot Study
Acronym: BREHAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Franciscus Gasthuis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-097
Record Dates: First submitted 2022-12-06; First posted 2023-10-11 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer; Lifestyle; Rehabilitation; Prehabilitation; Surgery
MeSH Terms: conditions — Breast Neoplasms | interventions — Preoperative Exercise; Rehabilitation

STUDY DESIGN:
Intervention Model Description: A pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prehabilitation/rehabilitation (Experimental): Patients in this arm follow a lifestyle counseling programme starting from diagnosis up to 6 months postoperatively.
  Interventions: Behavioral: Prehabilitation and rehabilitation
- Usual care (No Intervention): Patients in this arm follow usual care.

INTERVENTIONS:
Behavioral: Prehabilitation and rehabilitation — A personalized lifestyle counseling programme.
  Arms: Prehabilitation/rehabilitation

SUMMARY:
Prehabilitation and rehabilitation through personalized lifestyle counseling in patients with breast cancer.

ELIGIBILITY:
Inclusion criteria

1. Woman with a confirmed breast cancer diagnosis
2. Planned surgical treatment of breast cancer
3. Age 18 years or older
4. Provision of written informed consent

Exclusion criteria

1. Severe mental retardation, which limits the ability to follow instructions independently
2. Severe psychiatric problems, which limits the ability to follow instructions independently
3. Legal incapacity
4. Language barrier: If we cannot find a lifestyle coach who speaks the patient's language, unfortunately we cannot offer the lifestyle coaching in its entirety, and this option will be omitted for the patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Recruitment/consent rate | From baseline to 6 months postoperatively
  To estimate patient recruitment/consent rate to the prehabilitation/rehabilitation group Enrolment logs will be recorded for all patients who meet the eligibility criteria. Reasons for non-participation will be recorded. We define a success criterion of 40% of the total number of participants invited to be recruited to the pilot study.
Attendance rate | From baseline to 6 months postoperatively
  To estimate patient attendance, measured by the number of sessions attended out of 10. Reasons for non-attendance will be collected and withdrawals tracked. We will consider an attendance rate of 80% satisfactory
Patient adherence | From baseline to 6 months postoperatively
  To estimate patient adherence monitored with the aid of the wearables. Adherence is defined as at least 150 min of moderate intensity exercise and at least two strength training sessions per week. Exercise instructions are based on the Health Council's exercise guidelines. We will consider an adherence of 70% as satisfactory.
Withdrawals | From baseline to 6 months postoperatively
  To estimate the number of withdrawals, defined as the proportion of patients who quit the intervention before reaching the primary endpoint (HRQOL at six months after surgery). Information about the reasons for withdrawal will be collected.
Patient satisfaction | From baseline to 6 months postoperatively
  To estimate patient satisfaction with the programme assessed during three interviews: at four weeks, at three months after surgery and at the end of the study. Satisfaction is defined as: satisfaction with the lifestyle coach, satisfaction with the duration of the intervention, satisfaction with the physical training programme. Patients will be given room for their own input to improve the intervention.
Selection bias | From baseline to 6 months postoperatively
  To explore any evidence of selection bias in participants recruited into the study (assessed through participant characteristics at baseline).

SECONDARY OUTCOMES:
Likely changes in Health Related Quality of Life (HRQOL) | Baseline, the day before surgery, 6 months postoperatively
  To investigate likely changes in the primary outcome measure HRQOL measured with the EORTC-QLQ-30 questionnaire at six months after surgery.
Likely changes in BMI | Baseline, the day before surgery, 6 months postoperatively
  Body Mass Index
Likely changes in functional capacity (physical fitness) | Baseline, the day before surgery, 6 months postoperatively
  Measured using the 6 minute walking test (6MWT)
Likely changes in the number of postoperative complications | 30 days after surgery
  Complications within 30 days after surgery, measured with the Comprehensive Complication Index (CCI)
Likely changes in smoking status | Measured at baseline and 6 months postoperatively
  Smoking status (yes/no) as assessed by the primary investigator
Likely changes in postoperative functional recovery | The day after surgery
  Measured the day after surgery with the MILAS and DEMMI questionnaires
Likely changes in mean score of the different BREAST-Q scales | The questionnaire will be administered at enrolment and at six months after surgery.
  Measured using the BREAST-Q questionnaire
Likely changes in mean score of quality of life by means of the EORTC-BR23 questionnaire | The questionnaire will be administered at enrolment and at six months after surgery.
  Measured using the EORTC-BR23 questionnaire
Likely changes in mean score of the different EORTC-QLQ-30 scales which will be administered at enrolment and six months after surgery. | The questionnaire will be administered at enrolment and at six months after surgery.
  Measured using the EORTC-QLQ-30 questionnaire
Likely changes in mean score of the EQ5D-5L questionnaire | The questionnaire will be administered at enrolment and at six months after surgery.
  Measured using the EQ-5D-5L questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Taco Klem, MD,PHD, Principal Investigator — Franciscus Gasthuis & Vlietland
Locations (1):
- Franciscus Gasthuis en Vlietland, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No